CLINICAL TRIAL: NCT01923597
Title: A Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Effect of Green Tea on Albuminuria in Patients With Diabetic Nephropathy and Use of Maximum Dose of ACE-I and / or Angiotensin II Receptor Blocker.
Brief Title: Effect of Green Tea (Epigallocatechin Gallate) on Albuminuria in Patients With Diabetic Nephropathy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Cynthia de Moura Borges, master's student, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fapesp-2013
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2013-08

CONDITIONS: Diabetic Nephropathy; Hypertension
Keywords: Proteinuria; Oxidative stress; Epigallocatechin gallate
MeSH Terms: conditions — Diabetic Nephropathies; Hypertension; Proteinuria | interventions — Tea; epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Green tea extract (Active Comparator): Patients will receive four capsules ( one capsula = 200mg of epigallocatechin gallate) of green tea extract per day for 3 months.
  Interventions: Drug: Green tea extract
- Placebo (celulose) (Placebo Comparator): Patients will receive four capsules of placebo (celulose) daily for 3 months.
  Interventions: Drug: Green tea extract

INTERVENTIONS:
Drug: Green tea extract — 200mg/capsule Administered orally 4 capsules per day For 3 months
  Other Names: Epigallocatechin gallate; Polyphenol e

SUMMARY:
The purpose of this study is to determine the safety and effect of green tea (epigallocatechin gallate) in albuminuria in diabetic patients and nephropathy.

DETAILED DESCRIPTION:
Clinical, prospective, randomized, double-blind, placebo-controlled, with analysis by intention to treat.

50 individuals will be selected with a diagnosis of diabetes / hypertension and has been followed in Diabetic Nephropathy Clinic of the Faculty of Medical Sciences, University of Campinas (UNICAMP). Participants are divided into 02 groups: 1) 25 patients treated with maximum dose of ACE-I and / or angiotensin II receptor blocker (ARBs) + Placebo (absence of epigallocatechin gallate) and 2) treated 25 patients with maximum dose of ACE-I and / or ARBs + green tea (epigallocatechin gallate).

The patients will receive four capsules Polyphenol E - epigallocatechin gallate (Polyphenon Pharma, NY) per day, corresponding to 800 mg of epigallocatechin gallate (EGCG), or placebo (no epigallocatechin gallate) for 3 months. Patients will not be aware of the treatment they are receiving. The subjects will be allocated for the treatment or placebo, stratified by sex. To avoid the influence of researchers, the randomization list will be generated and maintained by trained personnel in a different location from the study. Before treatment and immediately after 3 months of treatment will be obtained in the primary outcome measures (albuminuria) and secondary (plasma metabolites of flavonoids, level of urinary F2-isoprostane and 8-hydroxydeoxyguanosine). In these same times will be obtained: blood biochemistry (glucose, glycosylated hemoglobin, urea, creatinine, sodium, potassium, blood count, calcium, phosphorus, cholesterol, LDL, HDL, triglycerides, uric acid), 3 samples of first morning urine to determine albuminuria, glomerular filtration rate (GFR), blood pressure measurement of 24 h, physical examination, weight, blood pressure and heart rate. Adherence to the study will be evaluated by weekly phone and the expected increase in plasma of flavonoids using the green tea (epigallocatechin gallate). The antihypertensive drug may be adjusted to obtain the desired pressure (<130/80 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* prior diagnosis of diabetes mellitus (DM)
* persistent micro-or macroalbuminuria (urinary albumin excretion> 30 mg / g creatinine (AUC) in 3 consecutive measurements on different days)
* glycated hemoglobin <10%
* maximum dose of ACE-I and / or ARBs.

Exclusion Criteria:

* diagnosis of autoimmune diseases, HIV, hepatitis, cancer, inflammatory disease
* pregnant or lactating patients
* glomerular filtration rate (GFR) <30 ml/min/1, 73m2 (estimated by the MDRD and the Cockcroft-Gault formula)
* presence of kidney disease unrelated to diabetes
* chronic urinary tract infection
* diagnosis of congestive heart failure (CHF) New York Heart Association (NYHA) class III or IV
* recent history (<6 months) unstable angina, myocardial infarction, stroke, coronary intervention
* history of alcohol and / or drugs
* mental incapacity to understand the informed consent
* intolerance to green tea

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effect of green tea (epigallocatechin gallate) in albuminuria in diabetic patients and nephropathy. | After 3 months of treatment
  Mean of 3 urinary albumin to creatinine ratio.

SECONDARY OUTCOMES:
Effect of green tea (epigallocatechin gallate) on oxidative stress in patients with diabetic nephropathy. | After 3 months of treatment
  Urinary levels of F2-isoprostane and 8-hydroxydeoxyguanosine
Effect of green tea (epigallocatechin gallate) on blood glucose control in patients with diabetic nephropathy. | After 3 months of tretatment
  Glycemia and glycated hemoglobin
Effect of green tea (epigallocatechin gallate) on blood pressure in patients with diabetic nephropathy. | After 3 months of treatment
  24 h blood pressure monitoring
Effect of green tea (epigallocatechin gallate) on plasma lipids in patients with diabetic nephropathy. | After 3 months of treatment
  Plasma levels of HDL.
Effect of green tea (epigallocatechin gallate) on plasma metabolites of flavonoids in patients with diabetic nephropathy. | After 3 months of treatment
  Plasma levels of epigallocatechin gallate and epicatechin.
Effect of green tea (epigallocatechin gallate) on plasma lipids in patients with diabetic nephropathy. | After 3 months of treatment
  Plasma levels of LDL.
Effect of green tea (epigallocatechin gallate) on plasma lipids in patients with diabetic nephropathy. | After 3 months of treatment
  Plasma levels of triglycerides.

OTHER OUTCOMES:
Effect of Green Tea (epigallocatechin gallate) in the glomerular filtration rate in patients with diabetic nephropathy. | After 3 months of treatment
  Estimated by Modification of Diet in Renal Disease (MDRD) formula.

CONTACTS AND LOCATIONS:
Overall Officials: José B. Lopes de Faria, MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Unicamp, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Faria AM, Papadimitriou A, Silva KC, Lopes de Faria JM, Lopes de Faria JB. Uncoupling endothelial nitric oxide synthase is ameliorated by green tea in experimental diabetes by re-establishing tetrahydrobiopterin levels. Diabetes. 2012 Jul;61(7):1838-47. doi: 10.2337/db11-1241. Epub 2012 May 14. PMID 22586583
- [Background] Ribaldo PD, Souza DS, Biswas SK, Block K, Lopes de Faria JM, Lopes de Faria JB. Green tea (Camellia sinensis) attenuates nephropathy by downregulating Nox4 NADPH oxidase in diabetic spontaneously hypertensive rats. J Nutr. 2009 Jan;139(1):96-100. doi: 10.3945/jn.108.095018. Epub 2008 Dec 3. PMID 19056645
- [Result] Borges CM, Papadimitriou A, Duarte DA, Lopes de Faria JM, Lopes de Faria JB. The use of green tea polyphenols for treating residual albuminuria in diabetic nephropathy: A double-blind randomised clinical trial. Sci Rep. 2016 Jun 20;6:28282. doi: 10.1038/srep28282. PMID 27320846
- See also: Results — http://www.nature.com/articles/srep28282